CLINICAL TRIAL: NCT06299254
Title: The Modulation of Individual Level of Fatigue Through Placebo Effect in Obesity
Brief Title: Placebo Effect About Fatigue in Obesity
Acronym: POF
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 21C305
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: placebo effect; fatigue; motivation; physical abilities
MeSH Terms: conditions — Obesity; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with obesity: Participants affected by obesity (the level of body mass index (BMI) higher or equal to 30).
  Interventions: Other: Placebo-Natural History
- Healthy-weight participants: As controls, not-hospitalized participants with a healthy weight
  Interventions: Other: Placebo-Natural History

INTERVENTIONS:
Other: Placebo-Natural History — Half of the participants will receive a placebo (i.e., motivational/verbal) cue before and after an experimental session in which they will perform several lifts.
  Half of the participants will receive no placebo before and after an experimental session in which they will perform several lifts.

SUMMARY:
Fatigue is a central symptom of obesity: it significantly impacts daily functioning, psychological well-being, compliance with physical therapy, and quality of life. However, the full understanding of the origin and treatment of fatigue in obesity is still a matter of debate, requiring further research, especially from new perspectives. From a neuroscientific perspective, fatigue is more than the subjective perception of tiredness resulting from mental or physical exertion or illness. It results in the complex interaction between (bottom-up) sensory input coming from the periphery, and motivational and psychological input, which is related to top-down cognition. In this framework, placebos may affect the output of the top-down cognitive processing by altering the individual evaluation of the ongoing peripheral performance. Indeed, evidence from both healthy conditions and clinical contexts suggests that fatigue can be modulated. The after-effect of such a modulation can be observed not only at a behavioural level, in terms of physical endurance, but also a psychological (i.e., decreased of perceived fatigue) and neurophysiological (changes in brain activity, especially in the fatigue-related components as the RP) levels.

ELIGIBILITY:
Inclusion criteria:

• Right-handed diagnosis of obesity (the level of body mass index - BMI - higher or equal to 30).

Exclusion criteria:

• concurrent neurological, neurodevelopmental (e.g., autism), motor, somatosensory and/or psychiatric disorders

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with obesity will be recruited at the beginning of a rehabilitative treatment at the Istituto Auxologico Italiano, IRCCS, San Giuseppe Hospital (Italy). Controls will be recruited out of the hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Behavioural outcome of fatigue | baseline
  The number of flexions (from a minimum of 0 to maximum of180) performed before and after the treatment for each individual.

SECONDARY OUTCOMES:
The individual level of perceived fatigue | baseline
  On a Likert scale (from 0 to 7), participants verbally report the individual level of perceived fatigue in doing the flexions before and after the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano - Ospedale San Giuseppe, Piancavallo, VCO, Italy